CLINICAL TRIAL: NCT03972306
Title: A Phase Ib, Open-Label, Multicenter Study To Investigate The Pharmacokinetics, Safety, And Tolerability Of Subcutaneous Ocrelizumab Administration In Patients With Multiple Sclerosis
Brief Title: A Study To Investigate The Pharmacokinetics, Safety, And Tolerability Of Subcutaneous Ocrelizumab Administration In Participants With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN41144
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: Cohorts A1-A4 (Experimental): Participants (participants pretreated with ocrelizumab) will receive a single injection of subcutaneous (SC) ocrelizumab co-mixed with rHuPH20 in the abdomen. For every new dose level, recruitment will be staggered by enrolling 1 participant in each cohort followed by a 48-hour waiting period to review safety and tolerability data by the Safety Monitoring Committee (SMC) prior to enrolling subsequent participants in the same cohort. Currently, the planned dose escalation steps for patients who enroll in Group A are as follows:
  * Cohort A1: 40 mg of SC ocrelizumab
  * Cohort A2: 200 mg of SC ocrelizumab
  * Cohort A3: 600 mg of SC ocrelizumab
  * Cohort A4: 1200 mg of SC ocrelizumab
  Interventions: Drug: Ocrelizumab; Drug: rHuPH20
- Group A: Cohort A5 (Experimental): In the non-randomized subphase, participants will receive a single SC injection of ocrelizumab co-mixed with rHuPH20 in the abdomen.
  Interventions: Drug: Ocrelizumab; Drug: rHuPH20
- Group A: Cohort AA (Experimental): Participants will receive a single 600-mg dose ocrelizumab by intravenous (IV) infusion
  Interventions: Drug: Ocrelizumab
- Group B: Cohorts B1-B4 (Experimental): Ocrelizumab treatment- naive participants will receive a minimum of 3 patients in Cohort B will receive a single SC injection of ocrelizumab co-mixed with rHuPH20 in the abdomen.
  * Cohort B1: 40 mg of SC ocrelizumab
  * Cohort B2: 200 mg of SC ocrelizumab
  * Cohort B3: 600 mg of SC ocrelizumab
  * Cohort B4: 1200 mg of SC ocrelizumab
  Interventions: Drug: Ocrelizumab; Drug: rHuPH20

INTERVENTIONS:
Drug: Ocrelizumab — Administered by subcutaneous Injection
  Arms: Group A: Cohort A5; Group A: Cohorts A1-A4; Group B: Cohorts B1-B4
Drug: Ocrelizumab — Administered by Intravenous (IV) Injection
  Arms: Group A: Cohort AA
Drug: rHuPH20 — Administered in a 2-mL glass vial as a sterile, single-use, injectable liquid to be manually mixed with SC ocrelizumab
  Arms: Group A: Cohort A5; Group A: Cohorts A1-A4; Group B: Cohorts B1-B4

SUMMARY:
This study will evaluate the pharmacokinetics, safety and tolerability, and immunogenicity of ocrelizumab administered subcutaneously to participants with multiple sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Progressive Multiple Sclerosis (PPMS) or Relapsing Multiple Sclerosis (RMS) according to the revised McDonald 2017 criteria (Thompson et al. 2018)
* Expanded Disability Status Scale (EDSS) score, 0-6.5, inclusive, at screening
* Absence of relapses for 30 days prior to the screening visit
* For the dose escalation phase for participants pretreated with ocrelizumab (Group A):

treatment with IV ocrelizumab for at least 1 year prior to screening (i.e., at least two 600-mg doses of ocrelizumab separated by 24 weeks)

* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods during the treatment period and for 6 months after the final dose of ocrelizumab.
* For female perticipants without reproductive potential:

Women may be enrolled if post-menopausal unless the participant is receiving a hormonal therapy for her menopause or if surgically sterile (i.e., hysterectomy, complete bilateral oophorectomy).

Exclusion Criteria:

* MS disease duration of more than 15 years for participants with an Expanded Disability Status Scale (EDSS) score <2.0 at screening.
* Known presence of other neurologic disorders that may mimic MS, including, but not limited to, the following:
* History of ischemic cerebrovascular disorders (e.g., stroke, transient ischemic attack) or ischemia of the spinal cord
* History or known presence of Central Nervous System (CNS) or spinal cord tumor (e.g., meningioma,glioma)
* History or known presence of potential metabolic causes of myelopathy (e.g., untreated vitamin B12 deficiency)
* History or known presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, human T-lymphotropic virus 1, herpes zoster and myelopathy.
* History of genetically inherited progressive CNS degenerative disorder (e.g., hereditary paraparesis and mitochondrial myopathy, encephalopathy, lactic acidosis, and stroke syndrome)
* Neuromyelitis optica
* History or known presence of systemic autoimmune disorders potentially causing progressive neurologic disease (e.g., lupus, anti-phospholipid antibody syndrome, Sjögren syndrome, Behçet disease, sarcoidosis).
* History of severe, clinically significant brain or spinal cord trauma (e.g., cerebral contusion, spinal cord compression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-Time Curve (AUC) of Ocrelizumab following subcutaneous (SC) administration | At predefined intervals from baseline through end of study (approximately 5 years)
Area Under the Serum Concentration-Time Curve (AUC) of Ocrelizumab following single IV (intravenous Infusion)administration | At predefined intervals from baseline through end of study (approximately 5 years)
Percentage of participants with adverse events | Baseline to end of study (approximately 5 years)
Percentage of participants with change from baseline in Marked Abnormality in Electrocardiogram (ECG) Parameters | Baseline to end of study (approximately 5 years)
Incidence of local pain at site of injection assessed using Visual Analog Scale (VAS | Baseline to end of study (approximately 5 years)
Incidence of local-injection reaction (ISR) assessed using Local Injection-Site Symptom Assessment (LISSA) | Baseline to end of study (approximately 5 years)

SECONDARY OUTCOMES:
Percentage of Participants with Anti-Drug Antibodies (ADAs) to ocrelizumab | Baseline to end of study (approximately 5 years)
Percentage of Participants with Anti-Drug Antibodies (ADAs) to rHuPH20 | Baseline to end of study (approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (18):
  - University of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The NeuroMedical Clinic of Central Louisiana, Alexandria, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Memorial Healthcare Institute for Neurosciences and Multiple Sclerosis, Owosso, Michigan
  - Washington Univ School of Med, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Mellen Center, Cleveland, Ohio
  - UC Health Neurology, Dayton, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Neurology Clinic PC, Cordova, Tennessee
  - University of Texas at Houston, Houston, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No